CLINICAL TRIAL: NCT00447304
Title: Acute Cholecystitis - Early Laparoscopic Surgery Versus Antibiotic Therapy and Delayed Elective Cholecystectomy = ACDC-study
Brief Title: Acute Cholecystitis - Early Laparoscopic Surgery Versus Antibiotic Therapy and Delayed Elective Cholecystectomy
Acronym: ACDC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-002056-14; AC-DC-01/Version 02/6.04.06
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2007-03

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis; cholecystectomy; antibiotic treatment; moxifloxacin; intraabdominal infection; morbidity and mortality of patients with acute cholecystitis, early surgery versus conservative therapy
MeSH Terms: conditions — Cholecystitis, Acute; Intraabdominal Infections | interventions — Moxifloxacin; Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: moxifloxacin
Procedure: cholecystectomy

SUMMARY:
Acute cholecystitis is frequent in the elderly, or in patients with gall stones. Most cases of severe or recurrent cholecystitis need surgery as final therapy. Today, the performed procedure in most cases for cholecystectomy in the western world is laparoscopic cholecystectomy. Only in some cases an open surgery has to be performed. Unclear is, what time point is best, concerning outcome and morbidity of the patient, immediate surgery or initial conservative therapy using antibiotics and symptomatic therapy with cholecystectomy later on. Today the performed procedure is mainly chosen by the fact, what doctor sees the patient first, surgeon or gastroenterologist. This study is performed to evaluate if one therapy is superior.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age > 18 years
* Patients with acute cholecystitis based on three of the following signs

  * abdominal pain in the upper right quadrant
  * Murphy's sign
  * leucocytosis > 10 /ml
  * rectal temperature > 38 °C or < 36.5 °C plus
  * cholecystolithiasis (stones / sludge) or sonographic signs of cholecystitis (thickening and triple layer formation of the gall bladder wall)
* Immediate antibiotic therapy (400 mg Moxifloxacin i.v. once a day)
* Laparoscopic cholecystectomy possible within 24 hours after presentation of the patient
* Informed consent

Exclusion Criteria:

* ASA IV and V (table 2)
* Septic shock
* Perforation or abscess of the gall bladder
* Impossibility of laparoscopic surgery (further surgery, surgeon, …)
* Additional need of antibiotics due to secondary disease
* Known intolerability of Moxifloxacin
* Known or possible pregnancy, breast feeding
* Life-threatening diseases (life-expectancy < 48 hours)
* End-stage liver disease (Child-Pugh C)
* Psychiatric or severe neurologic disease
* Relevant bradycardia or other symptomatic arrhythmias
* Significant cardiac disease
* Known long QT-disorders
* Electrolyte disorders, especially hypocalcemia
* Known intolerability of chinolones
* Earlier participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
morbidity at the test-of-cure visit

SECONDARY OUTCOMES:
Morbidity over 75 days using the score system showed in table 1
Morbidity 3 days after cholecystectomy (early or elective)
Necessity rate of conversion from laparoscopic to open surgery
Change of antibiotic due to non-response or non-toleration of moxifloxacin
Mortality at day 75
Cost-efficiency (comparing both trial branches)
Hospital time
Safety and tolerability of Moxifloxacin
In-hospital time after cholecystectomy (days)

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Buechler, Prof., Study Director — University Hospital Heidelberg, Department of Surgery, Heidelberg, Germany; Wolfgang Stremmel, Prof, Study Director — University Hospital Heidelberg, Department of Gastroenterology, Heidelberg, Germany
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Gutt CN, Encke J, Koninger J, Harnoss JC, Weigand K, Kipfmuller K, Schunter O, Gotze T, Golling MT, Menges M, Klar E, Feilhauer K, Zoller WG, Ridwelski K, Ackmann S, Baron A, Schon MR, Seitz HK, Daniel D, Stremmel W, Buchler MW. Acute cholecystitis: early versus delayed cholecystectomy, a multicenter randomized trial (ACDC study, NCT00447304). Ann Surg. 2013 Sep;258(3):385-93. doi: 10.1097/SLA.0b013e3182a1599b. PMID 24022431
- [Derived] Weigand K, Koninger J, Encke J, Buchler MW, Stremmel W, Gutt CN. Acute cholecystitis - early laparoskopic surgery versus antibiotic therapy and delayed elective cholecystectomy: ACDC-study. Trials. 2007 Oct 4;8:29. doi: 10.1186/1745-6215-8-29. PMID 17916243